CLINICAL TRIAL: NCT04081805
Title: LASER and Radiofrequency as Alternative Treatment of Vaginal Vulvar Atrophy in Women Treated for Breast Cancer
Brief Title: LASER and Radiofrequency for Treatment of Vaginal Vulvar Atrophy (VVA) in Women Treated for Breast Cancer (EPMLARF-arm2)
Acronym: EPMLARF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, Principal investigador, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP0431/2018 arm 2
Record Dates: First submitted 2019-08-08; First posted 2019-09-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Atrophy; Vulva; Atrophy; Breast Cancer
Keywords: LASER; Radiofrequency; Vulvovaginal atrophy; breast cancer; treatment
MeSH Terms: conditions — Atrophy; Breast Neoplasms | interventions — Lasers; Lasers, Gas; promestriene

STUDY DESIGN:
Intervention Model Description: The patient will be randomized in block to receive one of the three intravaginal therapies: LASER, Radiofrequency and promestriene
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcomes assessor will not have access to the treatment that was used in each patient.
  the investigator will not have acess to the treatment that was used in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LASER (Active Comparator): The patients will receive 3 consecutive applications of intravaginal and vulvar CO2 LASER, according to the manufacturer protocol for vaginal atrophy. The applications will be separated by the interval of 30 days
  Interventions: Procedure: LASER
- Micro Ablative Radiofrequency (Active Comparator): The patients will receive 3 consecutive applications of intravaginal and vulvar MIcroablative radiofrequency, according to the manufacturer protocol for vaginal atrophy. The applications will be separated by the interval of 30 days
  Interventions: Procedure: Micro Ablative Radiofrequency
- Promestriene (Active Comparator): The patient will use intravaginal promestriene, daily for 2 weeks and them twice a week for 3 months . Each 30 days, the patients will have an appointment when will be checked the weight of the promestriene tube to verify the correct use.
  Interventions: Drug: Promestriene

INTERVENTIONS:
Procedure: LASER — The patient will use intravaginal estriol, daily for 2 weeks and them twice a week for 3 months . Each 30 days, the patients will have an appointment when will be checked the weight of the estriol tube to verify the correct use.vulvar application of LASER, to postmenopausal genitourinary syndrome. The patient will be in gynecological position, after remove of vaginal secretion, with gauze and under topic anesthesia, the LASER will be applied, according to the protocol of the manufactured.
  Other Names: Fractional Co2 (carbon dioxide)Laser; MonaLisa Touch® treatment; SmartXide Touch V²LR® Deka
  Arms: LASER
Procedure: Micro Ablative Radiofrequency — Use of Linly™ equipment to perform ambulatory intravaginal and vulvar application of fractionated microablative radiofrequency, to postmenopausal genitourinary syndrome. The patient will be in gynecological position, after remove of vaginal secretion, with gauze and under topic anesthesia, the radiofrequency will be applied, according to the protocol of the manufactured
  Other Names: FRAAX; Linly™ Loktal Medical Electronics
  Arms: Micro Ablative Radiofrequency
Drug: Promestriene — The patient will perform self application of this vaginal promestriene daily for 2 weeks and after that the applications will occur twice a week.
  Other Names: Vaginal Promestriene
  Arms: Promestriene

SUMMARY:
This is a randomized controlled trial to evaluate the use of LASER, Micro Ablative radiofrequency and topic promestriene to treat symptoms of vulvovaginal atrophy of women treated for breast cancer.

DETAILED DESCRIPTION:
Women treated for breast cancer with moderate or severe signs or symptoms of vulvovaginal atrophy will be eligible for the study.

The patients will be randomized to receive one of the three intravaginal therapies: LASER, Micro Ablative radiofrequency or Promestriene. The applications will occur in the interval of 30 days for 3 times, for LASER and Radiofrequency groups. For the promestriene group, the application will be done by the patient, daily for 2 weeks and then twice a week for 3 months, and each 30 days, the patients will have an appointment when will be checked the weight of the promestriene tube, to verify the correct use.

The follow-up visits will occur 30, 90, 180 and 360 days after the conclusion of the third month of treatment.

Will be evaluated: vulvar and vaginal histology before and after the use of LASER, radiofrequency or estriol; microbiota and vaginal pH before and after the use of LASER, radiofrequency or promestriene; extracellular matrix and metalloproteinases in the remodeling of vulvovaginal collagen induced by promestriene, LASER and radiofrequency; quality of life, sexual dysfunctions and complains before and after the use of LASER, radiofrequency or hormones; metabolomics and vaginal microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Women with breast cancer treated with surgery and / or chemotherapy and / or radiotherapy, that has been concluded at least 6 months before inclusion, whether or not using aromatase inhibitor and complaining of vulvovaginal atrophy
2. To present, at least moderate, or severe intensity (score 4 or more of visual analog scale ( 0-10)) of one of the signs or symptoms of vulvovaginal atrophy:

   * Burning
   * Discomfort
   * Dryness
   * Cracks
   * Pruritus
   * Lack of vaginal lubrication
   * Penetration dyspareunia that began at the menopausal or postmenopausal transition
   * Decreased vaginal epithelium turgor and trophism
   * Deletion of mucous and skin folds.
3. Absence of vaginal surgical procedure in the last year
4. Genital prolapse stage no greater than stage II of Pelvic Organs Prolapse Quantitation (POP-Q) with Ba, Bp or C points less than or equal to 0

Exclusion Criteria:

1. Active genital infection
2. Active infection of HPV (human papillomavirus) or Herpes
3. users of medications with estrogenic effect (digoxin and other chemicals)
4. Postmenopausal genital bleeding
5. uncontrolled diabetes
6. use of multivitamins with zinc
7. use of copper or hormonal IUDs (intrauterine device) at the time of inclusion
8. presence of genitourinary or rectovaginal fistulas

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement of signs and symptoms of vulvovaginal atrophy with intravaginal LASER, Micro Ablative Radiofrequency, and topic promestriene | The evaluation will be done 90 days after treatment]
  Will be applied a Visual Analogic Scale (0-10) to access the improvement of genitourinary signs and symptoms, the results of the three groups will be compared
Satisfaction with treatment by intravaginal LASER, Micro ablative Radiofrequency, and topic promestriene for women treated for breast cancer, with genitourinary atrophy syndrome | The evaluation will be done 90 days after treatment
  Will be applied a LIKERT Satisfaction Scale (1-5) to access the satisfaction with the treatment, the results of the three groups will be compared

SECONDARY OUTCOMES:
Evaluation of Microbiota before and after the use of intravaginal LASER, Micro Ablative radiofrequency or topic promestriene | The evaluation will occur pre-treatment 30, 90 , 180 and 360 days after treatment]
  The vaginal flora will be evaluated by vaginal smear. The results of the three groups will be compared
Evaluation of vaginal pH before and after the use of intravaginal LASER, Micro ablative radiofrequency or topic promestriene | The evaluation will occur pre-treatment and 30, 90, 180 and 360 days after treatment
  The vaginal pH will be verified by the use of pH tape's. The results of the three groups will be compared
Histologic evaluation of vagina and vulva before and after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The evaluation will occur pre-treatment and 30 and 180 days after treatment
  Thickness of epithelium (mm and number of layers), and evaluation of expression of Ki-67 and VEGF (vascular endothelial growth factor) will be done on vaginal and vulvar biopsies, in order to evaluate the tissue regeneration ( a greater the number of layers associated with the expression of VEGF and ki67 indicate a tissue regeneration, the combination of this measures, and not evaluation each one isolated, are important to evaluate histological improvement). The results of the three groups will be compared
Evaluation of impact in Quality of life after treatment with intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The evaluation will occur pre-treatment and 30 and 180 and 360 days after treatment]
  The IQol (incontinence quality of life questionnaire, validated to portuguese language - score 0-100) will be used to evaluate quality of life .The results of the three groups will be compared
Evaluation of impact in Sexual function after treatment with intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The evaluation will occur pre-treatment and 30 180 and 360 days after treatment
  The FSF-I (Female Sexual Function Index , validated to portuguese language- score range from 2 - 36) will be used to evaluate sexual function . The results of the three groups will be compared
Evaluation of extracellular matrix before and after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The evaluation will occur pre-treatment and 30 and 180 days after treatment]
  Evaluation of the composition and concentration of the glycosaminoglycans of extracellular matrix in the vaginal and vulvar biopsies by specific markers. The results of the three groups will be compared
Evaluation of matrix metalloproteinases(MMP) in remodeling of vulvovaginal collagen induced by intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The evaluation will occur pre-treatment and 30 and 180 days after treatment
  Evaluation of the tissue distribution of the MMP-1, MMP-2, MMP-3, MMP-7, MMP-9 metalloproteinases of collagen I, II, IV and elastin proteins by specific markers on vaginal and vulvar biopsies. The results of the three groups will be compared
Evaluation of visual aspect of vulva after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic promestriene. | The pictures will be taken before and 30 days and 180 days after treatment.]
  Pictures of vulva will be taken before and after treatment. The images will be evaluated by a blind gynecologist and dermatologist regarding the type of treatment and the chronological order of the photos, which will classify the images as: better; equal or worse, in relation to tropism and number of vulvar skin grooves, The results of the three groups will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsanna IK Jarmy-di Bella, PhD, Study Chair — Professor; Marair GF Sartori, PhD, Study Director — Professor and Head of Gynecology Department
Locations (1):
- Federal University of Sao Paulo - Unifesp, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Cantarelli GC, Bianchi-Ferraro AMHM, Dedonatto C, Fernandes MFR, Vanzin RB, Dardes RCM, Logullo AF, de Almeida JS, Facina G, de Jarmy-Di Bella ZIK, Sartori MGF, Patriarca MT; LARF-Study Group. Clinical and histomorphometric evaluation of the vagina following treatment with CO2 laser, radiofrequency, and promestriene for genitourinary syndrome of menopause in breast cancer survivors on adjuvant therapy. Maturitas. 2025 Jan;191:108155. doi: 10.1016/j.maturitas.2024.108155. Epub 2024 Nov 14. PMID 39566128
- [Derived] Fernandes MFR, Bianchi-Ferraro AMHM, Sartori MGF, Jarmy Di Bella ZIK, Cantarelli GC, Dedonatto C, Vanzin RB, Dardes RCM, Logullo AF, Patriarca MT; LARF Study Group. CO 2 laser, radiofrequency, and promestriene in the treatment of genitourinary syndrome of menopause in breast cancer survivors: a histomorphometric evaluation of the vulvar vestibule. Menopause. 2023 Dec 1;30(12):1213-1220. doi: 10.1097/GME.0000000000002274. Epub 2023 Nov 14. PMID 37963315